CLINICAL TRIAL: NCT05523583
Title: Assessment of Tobacco Smoking and Alcohol Drinking and Treatment Outcomes Among Patients With Lung or Head and Neck Cancer
Acronym: SMALLHAN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0090
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lung or Head and Neck Cancer
Keywords: lung cancer; head and neck cancer; tabacco; alcohol
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms | interventions — Surveys and Questionnaires; Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients newly diagnosed with lung cancer or head & neck cancer: Patients newly diagnosed with lung cancer or head & neck cancer (International Classification of Diseases 10: C76, C34) who undergo front-line treatment and who had at least one episode of smoking within the past 30 days before diagnosis
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — A trained interviewer (Clinical Research Associate : CRA) will administer a questionnaire soon after the diagnosis on the phone (within 15 calendar days after diagnosis). The participants are followed up during the first year following the diagnosis through 3 follow-up assessments (at 3, 6, and 12 months after the baseline assessment) and hospital record reviews. At each follow-up, a brief questionnaire will be administered by an interviewer (CRA) via telephone.
  Other Names: Tabacco and alcohol questionnaires

SUMMARY:
The overarching goal of the proposed study is to provide information which can lead to effective implementation of cessation support in the care of smokers diagnosed with lung or head & neck cancer.

To achieve these aims, the study propose to conduct a longitudinal cohort study of patients diagnosed with lung or head & neck cancer at the Hospices Civils de Lyon (SMALLHAN). Briefly, adult patients newly diagnosed with lung or head & neck cancer will be recruited at the time of diagnosis (announcement of diagnosis and consultation).

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with lung cancer or head & neck cancer (International Classification of Diseases 10: C76, C34)
* Patients who undergo front-line treatment
* Age 18 years or older
* Benefiting from a Social Security scheme
* Written information about the study provided to the patient before any procedure specific to the study
* Patients who had at least one episode of smoking within the past 30 days before diagnosis

Exclusion Criteria:

* History of another lung or head & neck cancer < 5 years (Note: The presence of a second tumour location, discovered at the same time as the lung or head and neck cancer, does not constitute a non-inclusion criterion)
* History of another cancer (except for curatively treated cervical cancer in situ and non-melanoma skin cancer) < 3 years
* Mesothelioma, thymic malignancies, and cancer of the upper oesophagus
* Inability to complete the study for psychosocial reasons (inability to schedule interview (homeless), no access to phone, psychological disorder leading to inability to answer phone interview, do not speak French and no easy access to translator from surroundings)
* Patient under guardianship
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: .): Patients treated in HCL, newly diagnosed with lung cancer or head & neck cancer (International Classification of Diseases 10: C76, C34) who undergo front-line treatment and who had at least one episode of smoking within the past 30 days before diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Description of socio-professional determinants obtained by questionnaire | Baseline
  specific questionnaires querying demographics, socio-professional status, cessation or reduction attempts, and motivation and barriers to cessation, psychiatric conditions including level of addiction and depression.
Description of accessibility-related determinants obtained by questionnaire | Baseline
  specific questionnaire querying travel time, distance, means of transportation used to access the hospital or cessation services
Change of odds ratios and corresponding 95% confidence intervals for non-use of cessation services evaluated by questionnaire(0=non-use of service, 1=use of service) | Baseline and 3, 6 and 12 months
Change of odds ratios and corresponding 95% confidence intervals for continuation or relapse of tobacco use or dual use of tobacco and alcohol evaluated by questionnaire (0=abstinent, 1=continuation or relapse) | Baseline and 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Louis Pradel, Pneumologie, Bron
  - Hôpital de la Croix-Rousse, Oto-Rhino-Laryngologie et Chirurgie Cervico-Faciale, Lyon
  - Hôpital de la Croix-Rousse, Pneumologie, Lyon
  - Hôpital Lyon Sud, Pneumologie, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: Undecided
A decision on sharing individual participant data has not yet been made. Data sharing will depend on sponsor policy, ethical approval, and compliance with applicable regulations.